CLINICAL TRIAL: NCT04338542
Title: A Proof-of-concept Study Investigating the Comparison of the RAS Mutational Status Between Primary Tumor and Metastasis in Patients Affected by Metastatic Colorectal Cancer on the Basis of Different Chemotherapeutic Regimens
Brief Title: A Retrospective Study Project of Clinico-molecular Characterization in Patients With Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Sara De Dosso (Other)
Collaborators: Istituto Cantonale di Patologia (Other); Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Sara De Dosso, Department Senior, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Other Study IDs: IOSI-ICP-001
Record Dates: First submitted 2020-04-05; First posted 2020-04-08 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Mestastatic ColoRectal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- neoadjuvant chemotherapy plus bevacizumab: Patients treated with surgery of the primary tumor, neoadjuvant chemotherapy plus bevacizumab and, finally, the surgical resection of liver metastasis.
  Interventions: Genetic: Tumor biobsies analysis
- neoadjuvant chemotherapy: Patients treated with surgery of the primary tumor, neoadjuvant chemotherapy and, finally, the surgical resection of liver metastasis.
  Interventions: Genetic: Tumor biobsies analysis
- control group: Patients presenting with synchronous primary tumour and metastasis resected without any preoperative systemic therapy.
  Interventions: Genetic: Tumor biobsies analysis

INTERVENTIONS:
Genetic: Tumor biobsies analysis — Analysis on archived tumor biopsies

SUMMARY:
This is a retrospective, translational, proof-of-concept study on tumor biopsies done on patients affected by mCRC and exhibiting RAS mutation.

For each patient it will be selected the tissue biopsies of primary tumour and of paired resected metastasis.

DETAILED DESCRIPTION:
the study implies the subdivision into three groups with a 1:1:1 ratio.

* The first group includes patients treated with surgery of the primary tumor, neoadjuvant chemotherapy plus bevacizumab and, finally, the surgical resection of liver metastasis.
* The second group is similar to group one, with the exception that patients were not treated with a bevacizumab-based regimen.
* The third group, the control group, includes patients presenting with synchronous primary tumour and metastasis resected without any preoperative systemic therapy

Genomic DNA from formalin-fixed paraffin-embedded (FFPE) tissues from the primary tumor and metastatic lesions will be extracted. The genomic DNA will be assessed for the RAS mutational status in a quantitative and qualitative manner using two different approaches: a real-time PCR approach using the SensiScreen® kit (PentaBase Aps) and a next-generation sequencing approach using the Ion Torrent platform by applying the Ion AmpliSeq™ Cancer Hotspot Panel v2 (ThermoFisher Scientific). The real-time PCR is able to provide the relative quantification of the RAS mutant allele by comparing the Ct value of the mutation with respect to the Ct of the reference gene. This ratio will be calculated for both the primary tumor and for the metastasis and then compared. Ion Torrent gives directly the percentage of the mutant allele in each sample. Furthermore, the Cancer Hotspot Panel v2 provides data (both quantitative and qualitative) about the mutational status of additional 49 genes, including the most relevant and frequently mutated genes in CRC (i.e.: APC, TP53, PIK3CA, BRAF and PTEN) and the relative mutational pattern of the primary tumor and the one of the distant metastasis will be compared.

ELIGIBILITY:
General inclusion criteria (valid for all the three cohorts):

* patients with biopsy-proven, stage IV CRC;
* RAS mutation at diagnosis;
* availability of tissue biopsy/resection of both primary tumour and paired liver metastasis for the molecular characterization;

General exclusion criteria (valid for all the three cohorts):

* inadequate material for the molecular characterization of the primary tumour and/or of the related metastasis;
* insufficient amount (%) of tumour cells;

Specific inclusion criteria for each group:

1. st group:

   * first-line bevacizumab plus chemotherapy before resection of liver metastases;
   * metastases must be resected metachronously with respect to the primary tumor.
2. nd group:

   * first-line chemotherapy without bevacizumab before resection of liver metastases;
   * metastases must be resected metachronously with respect to the primary tumor.
3. rd group:

   * no systemic therapy (immediate surgical resection of primary tumor and paired liver metastases);
   * primary tumour and metastasis can be synchronous or metachronous.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: metastatic ColoRectal Cancer patients exhibiting RAS mutation and who received a treatment
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Change of RAS mutant clones in the metastatic lesion | 6 months
  To confirm that the administration of an antiangiogenic treatment in mCRC RAS mutant patients before liver metastasis resection leads to a significant reduction of RAS mutant clones in the metastatic lesion

SECONDARY OUTCOMES:
Molecular patterns other than RAS | 6 months
  Compare molecular patterns other than RAS in the primary tumor and paired liver metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Sara De Dosso, MD, Study Chair — Ente Ospedaliero Cantonale, Bellinzona; Milo Frattini, MD, Principal Investigator — Istituto Cantonale Patologia
Locations (1):
- Istituto Oncologico della Svizzera Italiana, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No